CLINICAL TRIAL: NCT06513091
Title: US National OCS Lung Thoracic Organ Perfusion (TOP) Registry
Brief Title: US National TOP Registry
Status: Recruiting | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCS-LUN-TOP-II
Record Dates: First submitted 2024-07-12; First posted 2024-07-22 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-02

CONDITIONS: Lung Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- OCS Lung Transplant Recipients: The US National TOP Registry will enroll all liver transplant recipients who are transplanted with OCS-perfused donor lung(s) in the Registry.
  Interventions: Device: OCS Lung
- Non-OCS Lung Transplant Recipients: Patients transplanted using other preservation modalities for benchmarking clinical outcomes.

INTERVENTIONS:
Device: OCS Lung — The TransMedics Organ Care System (OCS) Lung is an FDA approved portable extracorporeal lung perfusion and monitoring system.
  Groups: OCS Lung Transplant Recipients

SUMMARY:
The objective of this Registry is to collect short and long-term post-transplant clinical outcome data of all donor lungs preserved and assessed on the OCS Lung System and to document the performance of the OCS device in the real-world setting after FDA approval in the US.

ELIGIBILITY:
All lung transplant recipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The US National TOP Registry will enroll all lung transplant recipients who are transplanted with OCS-perfused donor lung(s) in the Registry, as well as patients transplanted using other preservation modalities for benchmarking clinical outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2034-11 (Estimated); Study Completion 2039-11 (Estimated)

PRIMARY OUTCOMES:
One-year patient and graft survival | 1-year post-transplant
  Recipients' one-year patient and graft survival rates

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Stanford University School of Medicine, Stanford, California
  - University of Minnesota, Minneapolis, Minnesota
  - Duke University, Durham, North Carolina
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin